CLINICAL TRIAL: NCT02909088
Title: An Open-label Study to Evaluate the Efficacy and Tolerability of Ecopipam in Adults With Childhood Onset Fluency Disorder (Stuttering).
Brief Title: Efficacy and Tolerability of Ecopipam in Adults With Childhood Onset Fluency Disorder (Stuttering).
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gerald Maguire, MD (Other)
Collaborators: University of California Riverisde School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Gerald Maguire, MD, Professor and Chair, Psychiatry and Neuroscience, Principal Investigator, CITrials
Organization: CITrials (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EcoUCR001; IND 128278 (Registry Identifier: FDA)
Record Dates: First submitted 2016-08-25; First posted 2016-09-21 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Stuttering, Adult; Childhood-onset Fluency Disorder; Speech Disorders; Language Disorders; Communication Disorder
Keywords: stuttering; childhood onset fluency disorder; ecopipam
MeSH Terms: conditions — Stuttering; Childhood-Onset Fluency Disorder; Speech Disorders; Language Disorders; Communication Disorders | interventions — ecopipam

ARMS (2):
- Ecopipam 50mg (Experimental): 50mg of ecopipam at bedtime for the first two weeks. If there is deemed improvement by the investigator, the subject will remain on the same dose. If there is no improvement, then the subjects' dose will be increased to 100mg at bedtime beginning on day 14.
  Interventions: Drug: Ecopipam 50mg; Drug: Ecopipam 100mg
- Ecopipam 100mg (Experimental): If there is no improvement, then the subjects' dose will be increased to 100mg at bedtime beginning on day 14.
  Interventions: Drug: Ecopipam 50mg; Drug: Ecopipam 100mg

INTERVENTIONS:
Drug: Ecopipam 50mg
Drug: Ecopipam 100mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy and tolerability of ecopipam in reducing stuttering symptoms.

It is hypothesized that ecopipam effectively reduces stuttering symptoms as measured on the SSI-IV total score, the CGI, SSS and OASES.

ELIGIBILITY:
Inclusion Criteria:

Subjects can be enrolled in the study only if they meet all of the following criteria:

1. Subjects must satisfy DSM-IV criteria for childhood onset fluency disorder (stuttering).
2. The nature of stuttering must be developmental in origin with the onset prior to ten years of age.
3. Subjects must have a score of moderate or higher on the SSI-IV.
4. Women of child-bearing potential are eligible to participate as long as they are practicing a medically accepted form of contraception (i.e. condom with spermicide or diaphragm, oral or depot contraception, or an intrauterine device).
5. Subjects will be male or female from the ages of 18-60.
6. Subject must have a MADRS total score of ≤ 13 (normal mood)
7. Subjects will be of only English speaking.

Exclusion Criteria:

Subjects will be excluded from the study for any of the following reasons:

1. Adult individuals who lack capacity to consent for themselves.
2. Stuttering related to a known neurologic cause (e.g. head trauma, stroke).
3. Unstable medical or psychiatric illness.
4. Active substance abuse within three months prior to study inclusion.
5. Any illness that would require the concomitant use of a CNS active medication during the course of the study.
6. Subjects with Parkinson's dementia or other degenerative neurologic illness.
7. Suffer from irregular heart rate or seizures
8. Subjects who are pregnant or nursing an infant.
9. Subject with a MADRS ≥ 14
10. Breastfeeding a child during the course of the study or for one month following completion
11. It is the investigator's opinion that the subject poses a significant suicide risk by the following criteria:

    1. It is the investigator's opinion that the subject may be at risk of suicide.
    2. the subject responds "yes" to question #4 (Active Suicidal Ideation with Specific Plan and Intent) on the Baseline Visit of the Columbia Suicide Severity Rating Scale (C-SSRS), if the most recent episode occurred within the past 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change in the Stuttering Severity Instrument Version IV (SSI-IV) | This scale is completed on Visit 1/screening and Visit 5/week 8.
  This is an objective measure of stuttering in which it captures verbal samples of five minutes speaking during a conversation and 5 minutes of reading a passage.

SECONDARY OUTCOMES:
Clinical Global Impression Scale-Severity (CGI-S) | This scale is completed on Visit 1/screening, Visit 2/baseline, Visit 3/week 2, and Visit 5/week 8.
  This is an evaluation of the patient by the investigator as to whether or not the subjects has improved, remained the same, or worsened while in the study.
Subjective Stuttering Scale (SSS) | This scale is completed on Visit 2/baseline and Visit 5/week 8.
Overall Assessment of the Speaker's Experience of Stuttering (OASES) | This scale is completed on Visit 2/baseline and Visit 5/week 8.
Montgomery Asberg Depression Rating Scale (MADRS) | This scale is completed on Visit 2/baseline, Visit 3/week 2, Visit 4/week 4 and Visit 5/week 8.
  An observer-rated depression scale
Barnes Akathisia Scale (BAS) | This scale is completed on Visit 1/screening, Visit 5/week 8.
  measures how restless the subject is during the examination
Abnormal Involuntary Movement Scale (AIMS) | This scale is completed on Visit 1/screening, Visit 5/week 8.
Columbia-Suicide Severity Rating Scale (C-SSRS) | This scale is completed on Visit 1/screening, Visit 2/baseline, Visit 3/week 2, Visit 4/week 4 and Visit 5/week 8.
Simpson Angus Scale (SAS) | This scale is completed on Visit 1/screening, Visit 5/week 8.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CITrials, Riverside, California
  - University of California Riverside School of Medicine, Riverside, California

REFERENCES:
- [Result] Maguire GA, Riley GD, Franklin DL, Maguire ME, Nguyen CT, Brojeni PH. Olanzapine in the treatment of developmental stuttering: a double-blind, placebo-controlled trial. Ann Clin Psychiatry. 2004 Apr-Jun;16(2):63-7. doi: 10.1080/10401230490452834. PMID 15328899
- [Result] Maguire GA, Yu BP, Franklin DL, Riley GD. Alleviating stuttering with pharmacological interventions. Expert Opin Pharmacother. 2004 Jul;5(7):1565-71. doi: 10.1517/14656566.5.7.1565. PMID 15212606
- [Result] Maguire G, Franklin D, Vatakis NG, Morgenshtern E, Denko T, Yaruss JS, Spotts C, Davis L, Davis A, Fox P, Soni P, Blomgren M, Silverman A, Riley G. Exploratory randomized clinical study of pagoclone in persistent developmental stuttering: the EXamining Pagoclone for peRsistent dEvelopmental Stuttering Study. J Clin Psychopharmacol. 2010 Feb;30(1):48-56. doi: 10.1097/JCP.0b013e3181caebbe. PMID 20075648
- [Result] Maguire GA, Riley GD, Yu BP. A neurological basis of stuttering? Lancet Neurol. 2002 Nov;1(7):407. doi: 10.1016/s1474-4422(02)00217-x. No abstract available. PMID 12849360
- [Result] Gilbert DL, Budman CL, Singer HS, Kurlan R, Chipkin RE. A D1 receptor antagonist, ecopipam, for treatment of tics in Tourette syndrome. Clin Neuropharmacol. 2014 Jan-Feb;37(1):26-30. doi: 10.1097/WNF.0000000000000017. PMID 24434529
- [Result] Riley J, Riley G, Maguire G. Subjective Screening of Stuttering severity, locus of control and avoidance: research edition. J Fluency Disord. 2004;29(1):51-62. doi: 10.1016/j.jfludis.2003.12.001. PMID 15026214
- [Result] Maguire GA, Riley GD, Franklin DL, Gottschalk LA. Risperidone for the treatment of stuttering. J Clin Psychopharmacol. 2000 Aug;20(4):479-82. doi: 10.1097/00004714-200008000-00013. PMID 10917410